CLINICAL TRIAL: NCT00907426
Title: Safety and Efficacy Study of Bimatoprost to Treat Hypotrichosis of the Eyelashes After Application to the Eyelid Margin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-038
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-08

CONDITIONS: Hypotrichosis
Keywords: eyelashes
MeSH Terms: conditions — Hypotrichosis | interventions — Bimatoprost; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bimatoprost 0.03% Followed by Bimatoprost 0.03% (Experimental): Treatment period one (0-6 months), once daily, one drop of Bimatoprost 0.03% solution using a single-use per eye applicator will be applied to the upper eyelid margin (where the eyelashes meet the skin). For treatment period two (6-12 months), once daily, one drop of Bimatoprost 0.03% solution using a single-use per eye applicator will be applied to the upper eyelid margin.
  Interventions: Drug: Bimatoprost 0.03% solution
- Bimatoprost 0.03% Followed by Vehicle (Other): Treatment period one (0-6 months), once daily, one drop of Bimatoprost 0.03% solution using a single-use per eye applicator will be applied to the upper eyelid margin (where the eyelashes meet the skin). For treatment period two (6-12 months), once daily, one drop of vehicle solution using a single-use per eye applicator will be applied to the upper eyelid margin.
  Interventions: Drug: Bimatoprost 0.03% solution; Drug: Vehicle solution
- Vehicle Followed by Bimatoprost 0.03% (Other): Treatment period one (0-6 months), once daily, one drop of vehicle solution using a single-use per eye applicator will be applied to the upper eyelid margin (where the eyelashes meet the skin). For treatment period two (6-12 months), once daily, one drop of Bimatoprost 0.03% solution using a single-use per eye applicator will be applied to the upper eyelid margin.
  Interventions: Drug: Bimatoprost 0.03% solution; Drug: Vehicle solution

INTERVENTIONS:
Drug: Bimatoprost 0.03% solution — Once daily, one drop of Bimatoprost 0.03% solution using a single-use per eye applicator will be applied to the upper eyelid margin (where the eyelashes meet the skin).
  Other Names: LATISSE™
Drug: Vehicle solution — Once daily, one drop of vehicle solution using a single-use per eye applicator will be applied to the upper eyelid margin (where the eyelashes meet the skin).
  Other Names: LATISSE™
  Arms: Bimatoprost 0.03% Followed by Vehicle; Vehicle Followed by Bimatoprost 0.03%

SUMMARY:
This one-year study evaluates the long-term safety and effectiveness of bimatoprost solution application to the eyelid margin (where the eyelashes meet the skin) to treat hypotrichosis of the eyelashes (inadequate or not enough eyelashes). There will be two different types of subjects participating in the study 1)those with inadequate eyelashes due to natural causes or 2) those with inadequate eyelashes following a complete course of chemotherapy treatment. There will be two treatment periods of six months each. Subjects will receive either the study medication or vehicle in either of the two treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have inadequate eyelashes due to natural causes and are not satisfied with their eyelash appearance.
* For the post-chemotherapy population: subjects who have inadequate eyelashes following a complete course of chemotherapy treatment and are not satisfied with their eyelash appearance, are considered free of cancer and are well enough to complete the study.

Exclusion Criteria:

* Subjects with unequal right and left eyelashes, any eye disease or abnormality, eye surgery, permanent eyeliner, eyelash implants, eyelash extension application.
* Any use of over the counter or prescription use eyelash growth products.
* Subjects requiring eye drop medications for glaucoma.
* Females who are pregnant, nursing or planning a pregnancy during the study or who are of childbearing potential and not using a reliable method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- San Diego, California, United States
- London, England, United Kingdom

REFERENCES:
- [Derived] Wirta D, Baumann L, Bruce S, Ahluwalia G, Weng E, Daniels S. Safety and Efficacy of Bimatoprost for Eyelash Growth in Postchemotherapy Subjects. J Clin Aesthet Dermatol. 2015 Apr;8(4):11-20. PMID 26060513
- [Derived] Harii K, Arase S, Tsuboi R, Weng E, Daniels S, VanDenburgh A. Bimatoprost for eyelash growth in Japanese subjects: two multicenter controlled studies. Aesthetic Plast Surg. 2014 Apr;38(2):451-60. doi: 10.1007/s00266-014-0293-7. Epub 2014 Mar 19. PMID 24643895

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1 (0 to 6 Months)
Arm/Group | Bimatoprost 0.03% Followed by Bimatoprost 0.03% | Bimatoprost 0.03% Followed by Vehicle | Vehicle Followed by Bimatoprost 0.03%
Started | 215 | 60 | 93
Completed | 195 | 55 | 84
Not Completed | 20 | 5 | 9
Period: Treatment Period 2 (6 to 12 Months)
Arm/Group | Bimatoprost 0.03% Followed by Bimatoprost 0.03% | Bimatoprost 0.03% Followed by Vehicle | Vehicle Followed by Bimatoprost 0.03%
Started | 195 | 55 | 84
Completed | 184 | 52 | 77
Not Completed | 11 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost 0.03% Followed by Bimatoprost 0.03% | Bimatoprost 0.03% Followed by Vehicle | Vehicle Followed by Bimatoprost 0.03% | Total
Number analyzed (Participants) | 215 | 60 | 93 | 368
Age, Customized [Number; unit: Participants]
  <45 Years | 56 | 18 | 31 | 105
  Between 45 and 65 years | 151 | 35 | 53 | 239
  >65 Years | 8 | 7 | 9 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 58 | 92 | 364
  Male | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Responders at Month 4
Description: Percentage of Treatment Responders at Month 4 defined by: a) at least a 1-grade improvement from baseline in the Global Eyelash Assessment (GEA) score, AND b) at least a 3-point improvement from baseline in the total score for Domain 2 of the Eyelash Symptom Questionnaire (ESQ). The GEA 4-point scale assessed eyelash prominence from 1 (minimal) to 4 (very marked). Domain 2 of the ESQ assessed subjective attributes of confidence, attractiveness, and professionalism rated on a 5-point scale from 1 (very much disagree) to 5 (very much agree) for a total score between 3 and 15.
Time Frame: Month 4
Population: Intent-to-Treat: All randomized subjects
Measure: Number; unit: Percentage of Subjects
Groups:
- Bimatoprost 0.03%: Once daily, one drop of Bimatoprost 0.03% solution using a single-use per eye applicator will be applied to the upper eyelid margin (where the eyelashes meet the skin).
- Vehicle: Once daily, one drop of vehicle solution using a single-use per eye applicator will be applied to the upper eyelid margin (where the eyelashes meet the skin).
Arm/Group | Bimatoprost 0.03% | Vehicle
Number analyzed (Participants) | 275 | 93
Percentage of Subjects | 39.3 | 10.9

2. Secondary Outcome: Change From Baseline in Upper Eyelash Length at Month 4
Description: Change from Baseline to in upper eyelash length at Month 4, measured in millimeters (mm). Data from both eyes were averaged for each subject for analysis. Changes from baseline represented by positive values indicated longer length, and changes from baseline represented by negative values indicated shorter length.
Time Frame: Baseline, Month 4
Population: Intent-to-Treat: All randomized subjects who had baseline and Month 4 data collected for this outcome measure
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | Bimatoprost 0.03% | Vehicle
Number analyzed (Participants) | 271 | 89
Millimeters (mm)
  Baseline | 5.40 (1.085) | 5.42 (1.138)
  Change from Baseline at Month 4 | 1.33 (1.110) | 0.07 (1.015)

3. Secondary Outcome: Change From Baseline in Average Progressive Upper Eyelash Thickness at Month 4
Description: Change from baseline in average progressive upper eyelash thickness at Month 4 was measured within 3 preset areas. Eyelash thickness was assessed across both eyes as an average of the 3 preset areas measured in millimeters squared (mm^2). Changes from baseline at Month 4 represented by positive values indicated increased eyelash thickness, and changes from baseline represented by negative values indicated thinner eyelash thickness.
Time Frame: Baseline, Month 4
Population: Intent-to-Treat: All randomized subjects who had baseline and Month 4 data collected for this outcome measure
Measure: Mean (Standard Deviation); unit: Millimeters squared (mm^2)
Arm/Group | Bimatoprost 0.03% | Vehicle
Number analyzed (Participants) | 216 | 71
Millimeters squared (mm^2)
  Baseline | 0.67 (0.376) | 0.82 (0.598)
  Change from Baseline at Month 4 | 0.59 (0.471) | -0.07 (0.520)

4. Secondary Outcome: Change From Baseline in Upper Eyelash Darkness at Month 4
Description: Change from baseline in upper eyelash darkness at Month 4 was determined by lash intensity within the spline (a narrow area approximately 5 pixels wide that bisects the area of interest). Upper eyelash darkness was measured in both eyes and averaged for analysis. Colors ranged from black=0 to white=255. Lower numbers on this continuum indicated darker colors. A negative number value change from baseline indicated increased eyelash darkening.
Time Frame: Baseline, Month 4
Population: Intent-to-Treat: All randomized subjects who had baseline and Month 4 data collected for this outcome measure
Measure: Mean (Standard Deviation); unit: Eyelash Intensity Units
Arm/Group | Bimatoprost 0.03% | Vehicle
Number analyzed (Participants) | 215 | 70
Eyelash Intensity Units
  Baseline | 151.36 (24.670) | 148.82 (26.445)
  Change from Baseline at Month 4 | -23.55 (20.787) | -2.60 (18.592)

5. Other Pre Specified Outcome: Percentage of Subjects With at Least a 1-Grade Improvement in Global Eyelash Assessment (GEA) Score at Month 4
Description: Percentage of subjects with at least a 1-grade improvement in GEA score at Month 4. The GEA scale is an investigator-graded 4-point scale of overall eyelash prominence where 1=minimal, 2=moderate, 3=marked, and 4=very marked prominence.
Time Frame: Month 4
Population: Intent-to-Treat: All randomized subjects who had baseline and Month 4 data collected for this outcome measure
Measure: Number; unit: Percentage of Participants
Arm/Group | Bimatoprost 0.03% | Vehicle
Number analyzed (Participants) | 275 | 92
Percentage of Participants | 73.8 | 28.3

ADVERSE EVENTS:
Description: The Safety Population included all subjects who received at least one dose of study medication and was used to analyze serious adverse events (SAEs) and adverse events (AEs). SAEs/AEs are reported by arm randomized, not by treatment received.
Arm/Group | Bimatoprost 0.03% Followed by Bimatoprost 0.03% | Bimatoprost 0.03% Followed by Vehicle | Vehicle Followed by Bimatoprost 0.03%
Serious Adverse Events (participants affected / at risk) | 20/214 | 3/60 | 9/92
Other Adverse Events (participants affected / at risk) | 75/214 | 21/60 | 36/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03% Followed by Bimatoprost 0.03% (N=214) | Bimatoprost 0.03% Followed by Vehicle (N=60) | Vehicle Followed by Bimatoprost 0.03% (N=92)
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 — Not related to study treatment
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0 | 0 — Not related to study treatment
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 | 0 | 0 — Not related to study treatment
Chest Pain (General disorders) | 0 | 1 | 0 — Not related to study treatment
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 — Not related to study treatment
Bronchitis (Infections and infestations) | 0 | 0 | 1 — Not related to study treatment
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Not related to study treatment
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Not related to study treatment
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Not related to study treatment
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 — Not related to study treatment
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Not related to study treatment
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Not related to study treatment
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Not related to study treatment
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 — Not related to study treatment
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Not related to study treatment
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Not related to study treatment
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 — Not related to study treatment
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 — Not related to study treatment
Lung Carcinoma Cell Type Unspecified Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — Not related to study treatment
Migraine (Nervous system disorders) | 1 | 0 | 0 — Not related to study treatment
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0 — Not related to study treatment
Vaginal Prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 — Not related to study treatment
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Not related to study treatment
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — Not related to study treatment
Breast Reconstruction (Surgical and medical procedures) | 1 | 0 | 1 — Not related to study treatment
Breast Cellulitis (Infections and infestations) | 0 | 0 | 1 — Not related to study treatment
Pneumonia (Infections and infestations) | 0 | 0 | 1 — Not related to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.03% Followed by Bimatoprost 0.03% (N=214) | Bimatoprost 0.03% Followed by Vehicle (N=60) | Vehicle Followed by Bimatoprost 0.03% (N=92)
Conjunctival Hyperaemia (Eye disorders) | 26 | 4 | 6
Punctate Keratitis (Eye disorders) | 12 | 3 | 5
Eyelids Pruritus (Eye disorders) | 10 | 4 | 5
Erythema of Eyelid (Eye disorders) | 9 | 6 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 0 | 5
Nasopharyngitis (Infections and infestations) | 5 | 4 | 4
Headache (Nervous system disorders) | 4 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo